CLINICAL TRIAL: NCT06750146
Title: French Prospective Study on Biliary Tract Drainage Guided by Endoscopic Ultrasound in Patients With Malignant Biliary Stenosis (RAINBOW)
Brief Title: Hot AXIOS™ for Bile Duct Drainage in Malignant Stenosis
Acronym: RAINBOW
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7209
Record Dates: First submitted 2024-12-02; First posted 2024-12-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Malignant Biliary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hot AXIOS™ Recipients (Experimental): The Hot AXIOS™ Stent is a flexible, fully covered self-expanding metal stent that is preloaded within the Electrocautery Enhanced Delivery System. Patients who meet all eligibility criteria will receive the Hot AXIOS™stent and their quality of life will be measured at baseline, two weeks after stent placement and two months after stent placement by the jaundice dimension of the EORTC QLQ-BIL21 questionnaire. A patient is considered enrolled after signing the study-specific Informed Consent Form (ICF). Patients who sign the ICF but subsequently do not meet one or more of the selection criteria will be considered screen failures and excluded from the study.
  Interventions: Device: Hot AXIOS™ Stent and Electrocautery Enhanced Delivery System

INTERVENTIONS:
Device: Hot AXIOS™ Stent and Electrocautery Enhanced Delivery System — The Hot AXIOS™ Stent and Electrocautery Enhanced Delivery System is commercially available and can be used to bridge two lumens or organs to create an internal drain, so as to drain the bile ducts in case of failure of ERCP.
  Other Names: Hot AXIOS™

SUMMARY:
The study is designed to highlight the effectiveness of the Hot AXIOS™ stent when used in accordance with standard medical practice on the evolution of the quality of life of patients with malignant biliary stenosis requiring drainage of the bile ducts after failure of ERCP, in the two months after stent placement.

DETAILED DESCRIPTION:
The study will evaluate the quality of life in patients with malignant biliary obstruction after the placement of a lumen-apposing metal stent via endoscopic ultrasound, with an emphasis on the improvement of quality of life measured as a reduction in jaundice. Improvement in jaundice is a direct indicator of effective bile drainage and is expected to correlate with an enhancement in overall quality of life. Quality of life will be measured by means of subject response to the EORTC QLQ-BIL21, a component of the European Organization for Research and Treatment of Cancer (EORTC) designed specifically to assess the quality of life in patients with biliary tract cancer. The QLQ-BIL21 consists of 21 questions which aim to evaluate specific symptoms and issues relevant to patients with biliary tract cancer, such as jaundice, pain, digestive problems and the psychosocial impact of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Willing and able to comply with study procedures and provide written informed consent
3. Patients with failed ERCP for treatment of suspected malignant biliary obstruction
4. Patients for whom an indication for Hot AXIOS™ stent placement has been determined

Exclusion Criteria:

1. Women who are pregnant, nursing or planning to become pregnant during the study
2. Patients with immediately resectable tumor or resectable during the two months of the study
3. Patients for whom the placement of a double pigtail prosthesis is planned by the investigator during the index procedure
4. Current participation in another investigation drug or device study that could interfere with the endpoints of this study
5. Persons under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Measurement - Jaundice Dimension | 2 months (± 15 days)
  The primary outcome is the difference between the measurement taken at 2 months of follow-up (± 15 days) and the baseline measurement of quality of life assessed by the jaundice dimension of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-BIL21). The QLQ-BIL21 consists of 21 questions to which respondents rate their experience with various symptoms or problems on a scale from 1 (Not at All) to 4 (Very Much); the jaundice dimension consists of three of those questions. A lower score correlates to fewer symptoms or problems.

SECONDARY OUTCOMES:
Quality of Life Measurement - Non-Jaundice Dimension | 2 months (± 15 days)
  The absolute difference between the measurement taken at 2 months of follow-up (± 15 days) and the baseline measurement of quality of life assessed by the non-jaundice dimension of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-BIL21). The QLQ-BIL21 consists of 21 questions to which respondents rate their experience with various symptoms or problems on a scale from 1 (Not at All) to 4 (Very Much); the non-jaundice dimension consists of 18 of those questions. A lower score correlates to fewer symptoms or problems.
Quality of Life Measurement - Global Score | 2 months (± 15 days)
  The absolute difference between the measurement taken at 2 months of follow-up (± 15 days) and the baseline measurement of quality of life assessed by the global score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-BIL21). The QLQ-BIL21 consists of 21 questions to which respondents rate their experience with various symptoms or problems on a scale from 1 (Not at All) to 4 (Very Much). A lower score correlates to fewer symptoms or problems.
Reduction in Bilirubin (Clinical Success) | 2 weeks (+ 7 days) and 2 months (± 15 days)
  Clinical success is defined as a reduction in bilirubin > 50% at each follow-up compared to baseline.
Rate of Resolution of Clinical Symptoms | 2 months (± 15 days)
  Resolution of GOO-related clinical symptoms such as jaundice, nausea/vomiting, fever/chills, weight loss and abdominal pain following implant of Hot AXIOS™ at 2 months of follow-up
Rate of Reintervention | 2 months (± 15 days)
  Reintervention is defined as endoscopic, radiological or surgical intervention for the management of recurrent biliary obstruction due to stent dysfunction (e.g., obstruction or migration) at 2 months of follow-up. This criterion will be measured within the population for whom the placement of the Hot AXIOS™ stent was a technical success.
Chemotherapy Status | 2 months (± 15 days)
  Number of days after study stent implantation to start or continuation of chemotherapy (if applicable).
Overall Survival | 2 months (± 15 days)
  Time from the placement of the Hot AXIOS™ to the date of death from any cause or to the end of follow-up (end of study participation or lost to follow-up) to assess summary measure overall survival.
Progression-Free Survival | 2 months (± 15 days)
  Time from the placement of the Hot AXIOS™ to the earliest date of either disease progression or death from any cause or to the end of follow-up (end of study participation or lost to follow-up) to assess summary measure progression-free survival.
Number of Days Alive after Hospital Discharge | 2 months (± 15 days)
  Number of days alive after hospital discharge within 2 months after the placement of the Hot AXIOS™.
Rate of Technical Success | 2 months (± 15 days)
  Technical success is defined as the successful placement of the Hot AXIOS™ stent during study procedure.
Serious Adverse Events | 2 months (± 15 days)
  Serious adverse events related to the study procedure and/or the Hot AXIOS™ stent.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Chevaux, Principal Investigator — Central Hospital, Nancy, France
Locations (18):
- France (18):
  - CHU de Besançon, Besançon
  - Clinique des Cedres, Ramsay Sante, Cornebarrieu
  - CHU Limoges, Limoges
  - Hopital Prive Jean Mermoz, Lyon
  - Clinique Jules Verne, Nantes
  - CHU Nice, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Paris Saint-Joseph, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - CHU de Poitiers, Poitiers
  - CHU Reims, Reims
  - CHRU Hopital Pontchaillou, Rennes
  - Clinique Saint-Hilaire, Rouen
  - Santé Atlantique, Saint-Herblain
  - CHU de Strasbourg, Strasbourg
  - CHU Rangueil, Toulouse
  - CHRU de Nancy, Vandœuvre-lès-Nancy
  - Centre Hospitalier de Vichy, Vichy

IPD SHARING:
Plan to Share IPD: No